CLINICAL TRIAL: NCT07212491
Title: Minimally Invasive Molecular Approaches for the Detection of Barrett's Esophagus- High Grade Dysplasia and Esophageal Adenocarcinoma- Renewal Grant Aim 2 (The SOS6C Trial)
Brief Title: Minimally Invasive Molecular Approaches for the Detection of Barrett's Esophagus- High Grade Dysplasia and Esophageal Adenocarcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: SOS6C; NCI-2025-06712 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-000761 (Other: Mayo Clinic Institutional Review Board); SOS6C (Other: Mayo Clinic Gastroenterology & Hepatology); R01CA241164 (NIH)
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained with permission of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo capsule sponge assessment over 5-10 minutes prior to standard of care endoscopy. Patients also undergo biopsy and esophageal brushing sample collection and complete questionnaires on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study explores the use of a minimally invasive screening tool (a sponge on a string device) to detect Barrett's esophagus and esophageal adenocarcinoma and to develop a laboratory test for the detection of Barrett's esophagus-high grade dysplasia and esophageal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient between the ages 18 - 90
* Patients with a BE segment >= 1cm in maximal extent endoscopically
* Histology showing evidence of intestinal metaplasia with or without presence of dysplasia
* Undergoing clinically indicated endoscopy

Exclusion Criteria:

* Patients with a prior history of ablation (photodynamic therapy, radiofrequency ablation, cryotherapy, argon plasma coagulation). Patients with a history of endoscopic mucosal resection alone will not be excluded
* Patients with a history of esophageal or gastric resection for esophageal or gastric carcinoma

  * Subjects with or without known evidence of BE (on history or review of medical records)
  * Pregnant or lactating females
  * Patients who are unable to consent
  * Patients with a current history of uninvestigated dysphagia (this does not apply to the brushings only portion of the study)
  * History of eosinophilic esophagitis, achalasia
  * Patients on oral anticoagulation including Coumadin, and warfarin, unless discontinued for five days prior to the sponge procedure
  * Patients on antiplatelet agents including clopidogrel, unless discontinued for five days prior to the sponge procedure
  * Patients on oral thrombin inhibitors including dabigatran and oral factor X an inhibitor such as rivaroxaban, apixaban, and edoxaban, unless discontinued for five days prior to the sponge procedure
  * Patients with a history of known varices or cirrhosis
  * Patients with a history of esophageal or gastric resection
  * Patients with congenital or acquired bleeding diatheses
  * Patients with a history of esophageal squamous dysplasia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a history of confirmed BE, undergoing clinically indicated endoscopy at Mayo Clinic Rochester, Mayo Clinic Florida, Mayo Clinic Arizona, Baylor Dallas, and University of Rochester, NY
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of deoxyribonucleic acid (DNA) markers | Baseline
  Will evaluate the sensitivity of DNA makers (methylated DNA markers ± aneuploidy) to distinguish between high-grade dysplasia (HGD)/esophageal adenocarcinoma (EAC) and non-dysplastic Barrett's esophagus (BE).
Specificity of DNA markers | Baseline
  Will evaluate the specificity of DNA markers (methylated DNA markers ± aneuploidy) to distinguish between HGD/EAC and non-dysplastic BE.

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G. Iyer, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials